CLINICAL TRIAL: NCT02742597
Title: Patient-Centred Innovations for Persons With Multimorbidity - Ontario
Acronym: PACEinMM-ON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other); Université de Sherbrooke (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Sunnybrook Health Sciences Centre (Other); Unity Health Toronto (Other); University Health Network, Toronto (Other); Michael Garron Hospital (Other); Providence Healthcare (Other); Mount Sinai Hospital, Canada (Other); Toronto Central Community Care Access Centre (Other); Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 104191
Record Dates: First submitted 2016-03-21; First posted 2016-04-19 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2020-09

CONDITIONS: Hypertension; Depression; Anxiety; Musculoskeletal Pain; Arthritis; Rheumatoid Arthritis; Osteoporosis; Chronic Obstructive Pulmonary Disease (COPD); Asthma; Chronic Bronchitis; Cardiovascular Disease; Heart Failure; Stroke; Transient Ischemic Attacks; Ulcer; Gastroesophageal Reflux; Irritable Bowel; Crohn's Disease; Ulcerative Colitis; Diverticulosis; Chronic Hepatitis; Diabetes; Thyroid Disorder; Cancer; Kidney Disease; Urinary Tract Problem; Dementia; Alzheimer's Disease; Hyperlipidemia; HIV; Multimorbidity
MeSH Terms: conditions — Hypertension; Depression; Anxiety Disorders; Musculoskeletal Pain; Arthritis; Arthritis, Rheumatoid; Osteoporosis; Pulmonary Disease, Chronic Obstructive; Asthma; Bronchitis, Chronic; Cardiovascular Diseases; Heart Failure; Stroke; Ischemic Attack, Transient; Ulcer; Gastroesophageal Reflux; Irritable Bowel Syndrome; Crohn Disease; Colitis, Ulcerative; Diverticulum; Hepatitis, Chronic; Diabetes Mellitus; Thyroid Diseases; Neoplasms; Kidney Diseases; Dementia; Alzheimer Disease; Hyperlipidemias | interventions — Lysine Acetyltransferase 5

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Active Comparator): Intervention group (n = 86) Intervention: Participates in Telemedicine Impact Plus (TIP)/ IMPACT Plus Care Coordination meeting
  Interventions: Behavioral: TIP / IMPACT Plus Care Coordination
- Group B (Active Comparator): Before/After Intervention group (n = 10) Intervention: Participates in TIP / IMPACT Plus Care Coordination meeting
  Interventions: Behavioral: TIP / IMPACT Plus Care Coordination
- Group C (No Intervention): Control group (n = 77)
- Group D (No Intervention): Health Administrative Data Group (n = 430) Number of matched data controls. Not taking part in intervention.

INTERVENTIONS:
Behavioral: TIP / IMPACT Plus Care Coordination — The intervention will involve the patient attending an interdisciplinary team meeting, either through the Ontario Telemedicine Network's teleconferencing technology or in person, along with their caregiver(s), the referring practitioner, inter-professional (IP) teams and home care coordinators to discuss and uncover the patient's condition covering a diverse range of medical, functional and psycho-social issues and the development of a patient-centred treatment plan. The care plans are documented, shared, implemented and monitored by an assigned nurse from the program.
  Arms: Group A; Group B

SUMMARY:
The aim of Patient-Centred Innovations for Persons With Multimorbidity (PACE in MM) study is to reorient the health care system from a single disease focus to a multimorbidity focus; centre on not only disease but also the patient in context; and realign the health care system from separate silos to coordinated collaborations in care. PACE in MM will propose multifaceted innovations in Chronic Disease Prevention and Management (CDPM) that will be grounded in current realities (i.e. Chronic Care Models including Self-Management Programs), that are linked to Primary Care (PC) reform efforts. The study will build on this firm foundation, will design and test promising innovations and will achieve transformation by creating structures to sustain relationships among researchers, decision-makers, practitioners, and patients. The Team will conduct inter-jurisdictional comparisons and is mainly a Quebec (QC) - Ontario (ON) collaboration with participation from 4 other provinces: British Columbia (BC); Manitoba (MB); Nova Scotia (NS); and New Brunswick (NB). The Team's objectives are: 1) to identify factors responsible for success or failure of current CDPM programs linked to the PC reform, by conducting a realist synthesis of their quantitative and qualitative evaluations; 2) to transform consenting CDPM programs identified in Objective 1, by aligning them to promising interventions on patient-centred care for multimorbidity patients, and to test these new innovations' in at least two jurisdictions and compare among jurisdictions; and 3) to foster the scaling-up of innovations informed by Objective 1 and tested/proven in Objective 2, and to conduct research on different approaches to scaling-up. This registration for Clinical Trials only pertains to Objective 2 of the study.

DETAILED DESCRIPTION:
A recent systematic review on the prevalence of Multimorbidity (MM) recommended a count of 3+ chronic diseases, with no focus on any single chronic disease in particular. This definition identifies a more vulnerable population with higher needs, lower income or poverty, poorer outcomes and challenging processes of care. It includes people with a wide array of complexity from the uncomplicated course of minimally interacting chronic diseases to the highly complex MM patients. MM is not only important due to the burden on patients, but because it accounts for high utilization. The definition represents a continuum of vulnerability in which there are many opportunities for prevention and management. Despite the high prevalence of MM, most research and health care is still based on a single disease paradigm which may not be appropriate as 45% of primary care patients have MM. A recent Cochrane systematic review on the impact of interventions for patients with MM has identified a paucity of studies internationally with mixed results, thus paving the way for the work of this Team. The most promising intervention, to date, was enhanced teamwork in a multifaceted intervention involving multiple professionals.

Patient-Centred Partnerships between Patients and Providers: The definition of patient-centred partnerships is derived from Canadian policy reports: "collaboration between informed, respected patients and a healthcare team." There is an internationally accepted comprehensive operational definition with four components which will guide many aspects of the proposed research program: first, exploring the patients' diseases and the illness experience; second, understanding the whole person in context; third, finding common ground; and fourth, enhancing the patient-provider relationship. There is empirical evidence for the impact of patient centred partnerships on better patient outcomes and lower costs. Systematic reviews of interventions indicated promising results for feasible practice-based interventions targeting both providers and patients.

Canadian policy reports defined this second facet of patient-centredness, as "seamless coordination and integration of care." Transitions requiring coordination are a key feature of care for patients with MM. Coordination has been shown to positively impact: symptom relief; social functioning; hospital re-admission and related costs. Papers reviewed by this Team identified the most promising type of intervention to be structured delivery system re-design.

STUDY #2.1 Qualitative Evaluation of the Aligned Programs Purpose: The study will: assess how the aligned program performs; distinguish between components of the interventions; and identify contextual factors that may have influenced the content and effectiveness of the intervention. It will also examine the local barriers and facilitators as well as the transitions and coordination of care.

Methods and design: The Team will conduct a qualitative evaluation of the aligned program to explain how various contexts influence observed effects [1] including the context of the health care systems in each province. A recent example of this research approach in Canada is Best et al, 2012 [2]. Data will be obtained from interviews and written documents. In-depth interviews will be conducted among the six categories of stakeholders. This will include: a) decision-makers (n = 10); b) providers (n = 10); c) family physicians and specialists (n = 10); d) a purposive sample of patients with multimorbidity (n = 10); e) family and informal caregivers (n=10); and f) referral providers (n = 10) [51]. Number of interviews are estimates and will be guided by the saturation of data [3].

Data collection: In-depth interviews, lasting 30 to 60 minutes will ensure complete and detailed participation. The data collection will be held during the second year of the transformed program. The interview guides will examine how the context variables influence the effects and the elements that could potentially inform the development of future interventions. All interviews will be audiotaped and transcribed verbatim. Additionally, written documents will be collected (program team meeting summaries, a sample of 10 medical records or research records at each participating site, a checklist describing the fidelity of the intervention, all documents produced specifically for the intervention) to provide an in-depth understanding of the various contexts in which the interventions occurred.

Data analysis: The data will be analyzed using an iterative and interpretative approach [4]. The data from all participants will be examined through both independent and team analysis occurring in a concurrent manner to build and develop on the emerging themes. A coding template will be developed and edited as new themes emerge while others are reclassified or discarded. The data management software NVivo 9.0 [QSR Int. USA] will be used to organize the coded data and identify exemplar quotes reflecting the central themes. All written documents will undergo a content analysis using NVivo 9.0. The final step of the analysis will be the triangulation of the synthesis of the themes from the stakeholder participants and the content analysis of the documents.[3-4] STUDY #2.2: Evaluation of effects of the Aligned Programs Setting: The same consenting participating sites as described in study 2.1. The methods presented below are for one setting and will be duplicated in the second setting. Patients are referred to receive the services of these programs by their providers. The intervention the investigators are testing here is the aligned programs. Patients referred to these programs are new patients and have never been exposed to the intervention. In addition to the main reason for referral to the program, the referral form will also include eligibility details for the evaluation, including diagnoses.

Patient sample: Patients recruited for the study will be cognitively intact and literate and aged between 18 and 80 years of age. The upper limit of 80 years is to avoid recruiting patients at risk of being institutionalized or dependent during the follow-up. Patients will present at least three chronic conditions.

Methods and Design: Patients agreeing to participate will complete questionnaires at baseline (T1) collecting the socio-demographic data and baseline measures, which will be used to document equivalence between groups (groups are defined below). Effectiveness of the aligned programs will be assessed using three strategies.

1. To measure short-term effects (4 months), a randomized controlled trial (RCT) design with a before/after arm will be used [5]. Eligible patients will be randomized after consent to receive either the intervention within a short period of time (Group A) or control (Group C); The before/after arm (Group B) will receive the intervention without being placed into the RCT, as their doctors have deemed them too fragile to risk randomization; Control participants (Group C) will receive a list of healthcare resources they may contact to assist with their care; questionnaires will be completed at baseline (T1), and 4 months post enrollment (Group C) or intervention (Group A & B) (T2) for all study participants. This will constitute the short-term measure of effectiveness of the intervention.
2. To measure the mid-term effects, the study participants will complete the same questionnaire 16 months post-enrollment (Group C) or intervention (Group A & B) (T3).
3. To measure mid-term (T3) and long-term effects (T4 after 2 years) on health services utilization and cost, study participants in Groups A and B will provide consent to give access to their health administrative (HA) data. A control Group D will be constituted using anonymized HA data. Patients will be matched for gender, age, region and three main diagnoses. The Team will build algorithms for matching every set of controls. Groups A and B together will be compared to this propensity matched control Group D using administrative (HA) data.

Variables and outcome measures: The variables fall into 5 categories: sociodemographic; PC context; main covariables of interest; primary outcomes; secondary outcomes. Sociodemographic characteristics include gender, age, education, family income, marital status, occupation, housing and number of persons living under the same roof. Context variables refer to type of PC organization in which the intervention occurs (solo or group practices, Family Health Team, Community Health Centre). The three main covariables of interest are the Team's three innovations: self-reported multimorbidity (measured by the Disease Burden Morbidity Assessment [6]; patient-centred partnership (Patient Perception of Patient-Centredness Scale [7-9]); and Patient centered coordination (the Patient Perceptions of Transitions in care, adapted by the investigators from Coleman [10]). The two primary outcome measures are the Health Education Impact Questionnaire (HeiQ) that provides a broad profile of the potential impacts of patient education interventions [11] and the level of perceived disease-management self-efficacy using the 6-item Self-Efficacy for Managing Chronic Disease (SEM-CD) [12]. Secondary patient perceived outcomes will be the VR-12 as a measure of health status and the EQ5D as a measure of Quality of Life [13]. The Kessler psychological distress scale K-6 will measure psychological distress [14]. The investigators will also use a questionnaire on health behaviors [15]. Finally, HA data will also be used as secondary outcomes to compare health care utilization and cost before and after the intervention. HA data will include emergency department visits, avoidable hospital admissions, readmissions, time to first primary care visit after emergency department visit and continuity of care.

Data analysis: The investigators will first describe participants' baseline characteristics in each group and compare among groups. To evaluate short-term effect, Groups A and C will be compared on T2 scores with an analysis of covariance (ANCOVA) adjusted for T1 scores [16]. To document mid-term effects, a before/after analysis of variance will be used to study the evolution of continuous variables collected 3 times [17]. Sub-analyses by gender will be performed. Health system costs in intervention and control groups will be evaluated by using amounts paid to providers based on provincial fee schedules and cost-weighted utilization of institutions including hospitals and long-term care. Utilization records obtained from HA data will be multiplied by applicable cost weights (e.g. CIHI Resource Intensity Weights - RIWs) and using CIHI costs per weighted case [18] The methods employed will model the individual patient-level costs incurred in the health system, using methods developed for costing using administrative data[19]. Incremental resources in the intervention group will be identified and costed using applicable time/resource inputs and relevant wage rates following guidelines for economic evaluation in health interventions [20].

ELIGIBILITY:
For Quantitative (Study 2.2):

Inclusion Criteria for Patients:

* 3+ Chronic Conditions
* 18 to 80 years of age
* Eligible for TIP/IMPACT Plus program
* Must live in catchment area for TIP/IMPACT Plus program (Toronto, Ontario, Canada)

Exclusion Criteria for Patients:

* Unable to reasonably respond to questionnaires or provide informed consent (ie. cognitive impairment or language barrier)
* Deemed by provider to be too fragile

For Qualitative (Study 2.1):

Inclusion Criteria:

* Decision Makers: Responsible for policy and financial decisions related to the TIP / IMPACT Plus program
* TIP / IMPACT Providers: Providers that have delivered the TIP / IMPACT Plus intervention to at least one patient, including pharmacist, nurse, nurse practitioner, physiotherapist, social worker, dietitian, occupational therapist, personal care worker / home care coordinator
* Family Physicians / Specialists: Those that take part in the TIP / IMPACT Plus intervention, including internist, psychiatrist, and family physician
* Patients: Need to meet the inclusion criteria of the TIP / IMPACT Plus program, 18 to 80 years of age, 3+ chronic conditions, and have received the intervention a minimum of 4 months prior to the qualitative interview
* Family and Caregivers: Need to be a family member or caregiver of a TIP / IMPACT Plus patient that has received the intervention a minimum of 4 months prior to the qualitative interview.
* Referral Provider: Emergency Department doctor, nurse practitioner, CCAC coordinator or representative community family doctor that has referred patients to the TIP / IMPACT Plus program.

Exclusion criteria:

* Decision Makers that are not knowledgeable about or involved with the TIP / IMPACT Plus program
* Providers/Family Physicians/Specialists that have not ever referred to or taken part in a TIP / IMPACT Plus intervention or have not been active with the program in the last year
* Family and Caregivers of Patients or Patients themselves that haven't yet received the TIP / IMPACT Plus intervention or those that received the intervention within the last 4 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2019-04-07 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of Intervention Effectiveness - Change in Self-Management outcomes | T1: Initial evaluation; T2: after 4 months; T3: one year after T2;
  Health Education Impact Questionnaire (HeiQ). Score: Reliable improvement
Evaluation of Intervention Effectiveness - Change in Transitions of Care | T1: Initial evaluation; T2: after 4 months; T3: one year after T2;
  Patient Perception of Transitions of Care. Score: Mean
Evaluation of Intervention Effectiveness - Change in Self-Efficacy | T1: Initial evaluation; T2: after 4 months; T3: one year after T2;
  Self-Efficacy for Managing Chronic Disease Scale (SEM-CD). Score: Mean
Evaluation of Intervention Effectiveness - Change in Patient-Centredness | T1: Initial evaluation; T2: after 4 months; T3: one year after T2;
  Patient Perception of Patient-Centredness (PPPC). Score: Mean

SECONDARY OUTCOMES:
Evaluation of Intervention Effectiveness - Change in Chronic Diseases | T1: Initial evaluation; T2: after 4 months; T3: one year after T2;
  Multimorbidity/Chronic Disease (MM-21): Score: Number of Chronic diseases
Evaluation of Intervention Effectiveness - Change in Health Status | T1: Initial evaluation; T2: after 4 months; T3: one year after T2;
  Health Status (VR-12): Score: Physical Component Summary (PCS) and the Mental Component Summary (MCS)
Evaluation of Intervention Effectiveness - Change in Quality of Life | T1: Initial evaluation; T2: after 4 months; T3: one year after T2;
  Quality of Life (EQ-5D-5L): Score: Mean
Evaluation of Intervention Effectiveness - Change in Psychological Well-being | T1: Initial evaluation; T2: after 4 months; T3: one year after T2;
  Psychological Well-being (Kessler 6 Scale). Score: Mean
Evaluation of Intervention Effectiveness - Change in Lifestyle/Health Behaviours | T1: Initial evaluation; T2: after 4 months; T3: one year after T2;
  Lifestyle/Health Behaviours Questionnaire. Score: Mean
Evaluation of Intervention Effectiveness - Change in Equity | T1: Initial evaluation; T2: after 4 months; T3: one year after T2;
  Vertical Equity. Score: Mean
Evaluation of Intervention Effectiveness - Change in Demographics | T1: Initial evaluation; T2: after 4 months; T3: one year after T2;
  Demographics. Score: frequencies, means

CONTACTS AND LOCATIONS:
Overall Officials: Moira Stewart, Principal Investigator — Western University
Locations (9):
- Canada (9):
  - Western University, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Providence Healthcare, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Central Community Care Access Centre, Toronto, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - University Hospital Network, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
De-identified subsets of data will be transferred upon request to healthcare providers at collaborating institutions under separate ethics approvals as/if required. Any transfers will be conducted by secure file transfer between encrypted devices. Any health information transferred will be de-identified.
Supporting Information: Study Protocol, CSR
Time Frame: Study Protocol: 2017 onward Clinical Study Report: 2020 onward
Access Criteria: The study protocol is available in a published paper (CMAJ Open 2017) Clinical Study Report: results published in British Journal of General Practice 2020

REFERENCES:
- [Background] Best A, Greenhalgh T, Lewis S, Saul JE, Carroll S, Bitz J. Large-system transformation in health care: a realist review. Milbank Q. 2012 Sep;90(3):421-56. doi: 10.1111/j.1468-0009.2012.00670.x. PMID 22985277
- [Background] Pawson, R. and N. Tilley, Realistic evaluation. London: Sage Publications Inc., 1997.
- [Background] Patton, M.Q., Qualitative Research & Evaluation. 3rd ed. Thousand Oaks, CA: Sage Publications Inc., 2002.
- [Background] Crabtree, B.F. and W.L. Miller, Doing Qualitative Research. Thousand Oaks, CA: Sage Publications Inc., 1999.
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; Consolidated Standards of Reporting Trials Group. CONSORT 2010 Explanation and Elaboration: Updated guidelines for reporting parallel group randomised trials. J Clin Epidemiol. 2010 Aug;63(8):e1-37. doi: 10.1016/j.jclinepi.2010.03.004. Epub 2010 Mar 25. PMID 20346624
- [Background] Poitras ME, Fortin M, Hudon C, Haggerty J, Almirall J. Validation of the disease burden morbidity assessment by self-report in a French-speaking population. BMC Health Serv Res. 2012 Feb 14;12:35. doi: 10.1186/1472-6963-12-35. PMID 22333434
- [Background] Stewart M, Brown JB, Donner A, McWhinney IR, Oates J, Weston WW, Jordan J. The impact of patient-centered care on outcomes. J Fam Pract. 2000 Sep;49(9):796-804. PMID 11032203
- [Background] Stewart M, Brown JB, Hammerton J, Donner A, Gavin A, Holliday RL, Whelan T, Leslie K, Cohen I, Weston W, Freeman T. Improving communication between doctors and breast cancer patients. Ann Fam Med. 2007 Sep-Oct;5(5):387-94. doi: 10.1370/afm.721. PMID 17893379
- [Background] Stewart, M., et al., The patient perception of patient-centeredness questionnaire (PPPC). Working Paper Series #04-1, April 2004.
- [Background] Coleman EA, Mahoney E, Parry C. Assessing the quality of preparation for posthospital care from the patient's perspective: the care transitions measure. Med Care. 2005 Mar;43(3):246-55. doi: 10.1097/00005650-200503000-00007. PMID 15725981
- [Background] Nolte S, Elsworth GR, Sinclair AJ, Osborne RH. The extent and breadth of benefits from participating in chronic disease self-management courses: a national patient-reported outcomes survey. Patient Educ Couns. 2007 Mar;65(3):351-60. doi: 10.1016/j.pec.2006.08.016. Epub 2006 Oct 5. PMID 17027221
- [Background] Sherer, M., et al., The self-efficacy scale: Construction and validation. Psychological Reports. 51: p. 663-671, 1982.
- [Background] Rasanen P, Roine E, Sintonen H, Semberg-Konttinen V, Ryynanen OP, Roine R. Use of quality-adjusted life years for the estimation of effectiveness of health care: A systematic literature review. Int J Technol Assess Health Care. 2006 Spring;22(2):235-41. doi: 10.1017/S0266462306051051. PMID 16571199
- [Background] Kessler RC, Barker PR, Colpe LJ, Epstein JF, Gfroerer JC, Hiripi E, Howes MJ, Normand SL, Manderscheid RW, Walters EE, Zaslavsky AM. Screening for serious mental illness in the general population. Arch Gen Psychiatry. 2003 Feb;60(2):184-9. doi: 10.1001/archpsyc.60.2.184. PMID 12578436
- [Background] Centers for Disease Control and Prevention (CDC), Behavioral Risk Factor Surveillance System Survey Questionnaire. 2007, Atlanta, Georgia: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention.
- [Background] Van Breukelen GJ. ANCOVA versus change from baseline: more power in randomized studies, more bias in nonrandomized studies [corrected]. J Clin Epidemiol. 2006 Sep;59(9):920-5. doi: 10.1016/j.jclinepi.2006.02.007. Epub 2006 Jun 23. PMID 16895814
- [Background] Daniel, W.W., Biostatistics: A foundation for analysis in the health sciences. 9th ed. Hoboken, NJ: Wiley, 2009.
- [Background] Canadian Institute for Health Information. Canadian Hospital Reporting Project (CHRP). 2012; https://secure.cihi.ca/free_products/HI2013_Jan30_EN.pdf . Accessed March 14, 2016.
- [Background] Wodchis, W.P., et al., Guidelines on Person-Level Costing Using Administrative Databases in Ontario. Toronto: Health System Performance Research Network, 2011.
- [Background] Drummond, M.F., et al., Methods for the economic evaluation of health care programmes. 3rd ed. New York: Oxford University Press, 2005.
- [Derived] Stewart M, Fortin M; Patient-Centred Innovations for Persons with Multimorbidity Team*. Patient-Centred Innovations for Persons with Multimorbidity: funded evaluation protocol. CMAJ Open. 2017 May 9;5(2):E365-E372. doi: 10.9778/cmajo.20160097. PMID 28487349
- See also: Website for PACE in MM — http://www.paceinmm.recherche.usherbrooke.ca/